CLINICAL TRIAL: NCT03727542
Title: Influence of Short AV Delay Pacing on Matrix Metalloproteinase Lives
Brief Title: Influence of Short AV Delay Permanent Pacing on Matrix Metalloproteinase Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr. Murat Sezer, Clinical Professor, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IU-1140
Record Dates: First submitted 2018-10-28; First posted 2018-11-01 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Aortic Aneurysm; Aortic Diseases; Pacemaker DDD
MeSH Terms: conditions — Aortic Aneurysm; Aortic Diseases

STUDY DESIGN:
Intervention Model Description: Serum level of MMP-9 will be measured initially in the blood samples collected from the patients with permanent pacemaker implantation while they were on sinus rhythm and the second samples will be collected at the end of the 3 weeks of short AVD (60 msec. shorter than patients' native PR interval) pacing to ensure wide QRS rhythm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Short AV-delay pacing (Experimental): Participants will be their own control. Serum samples will be collected at baseline while the participants were in sinus rhythm and after 3 weeks of short AV-delay pacing serum samples will be recollected to measure matrix metalloproteinase levels .
  Interventions: Device: adjustment of atrioventricular delay in DDD packers

INTERVENTIONS:
Device: adjustment of atrioventricular delay in DDD packers — Atrioventricular delays are going to be adjusted as 60 milisecond shorter than the patients' native PR intervals in patients with already implanted permanent pacemakers.

SUMMARY:
As potential biomarkers of pressure-related aortic damage, matrix metalloproteinases (MMP) have been implicated in the pathogenesis of aortic aneurysm because of the important role they play in connective tissue homeostasis. In particular, a significant reduction in initially elevated serum MMP - 9 concentrations, compared with healthy controls, demonstrated after the aortic repair in patients with abdominal aortic aneurysm implies MMPs pivotal role in aortic aneurysms. Besides, due to an active degradation and repair processes taking place in the vascular wall governed by the balance between MMP enzymes and their inhibitors, MMP - 9, expression of which is predominantly associated with disruption of aortic elastic fibers, can also be detected in the serum of healthy subjects. Indeed, mechanical stress-induced upregulation of genes and their products stimulate MMP expression in the vascular wall, which is responsible for extracellular matrix degradation. Herein, it was hypothesized that reducing the acceleration rate of aortic pressure (aortic peak dP/dt) may decrease the mechanical stretch on the aortic wall which, may in turn, reduce the expression and serum levels of MMP-9.

DETAILED DESCRIPTION:
The maximum value of acceleration rate of aortic pressure rise can be named as aortic peak dP/dt. It, likewise, corresponds to the maximum value of first derivative of aortic pressure curve with respect to time.Notably, aortic peak dP/dt would be one of the principal determinants of mechanical stress applied to the aortic wall. Hence, interventions aiming to reduce aortic peak dP/dt levels may open a new therapeutic avenue in the management of pressure-related vascular damages such as aortic aneurisms.

Since it is the principle determining factor of aortic peak dP/dt, changing LV contractility, thereby LV peak dP/dt, may be expected to lead to change aortic peak dP/dt values in the same direction. Therefore, reduction of LV dP/dt can lead to a reduction in aortic dP/dt. Previous finding strongly suggest that widening of the QRS complex could decrease LV contractility and correspondingly LV peak dP/dt value which may eventually lead to a reduction in aortic peak dP/dt.

From biomechanical point of view, as potential biomarkers of pressure-related aortic damage, matrix metalloproteinases (MMP) have been implicated in the pathogenesis of aortic aneurysm because of the important role they play in connective tissue homeostasis. In particular, a significant reduction in initially elevated serum MMP - 9 concentrations, compared with healthy controls, demonstrated after the aortic repair in patients with abdominal aortic aneurysm implies MMPs pivotal role in aortic aneurysms. Besides, due to an active degradation and repair processes taking place in the vascular wall governed by the balance between MMP enzymes and their inhibitors, MMP - 9, expression of which is predominantly associated with disruption of aortic elastic fibers, can also be detected in the serum of healthy subjects. Indeed, mechanical stress-induced upregulation of genes and their products stimulate MMP expression in the vascular wall, which is responsible for extracellular matrix degradation. Herein, we hypothesized that reducing the acceleration rate of aortic pressure (aortic peak dP/dt) may decrease the mechanical stretch on the aortic wall which, may in turn, reduce the expression and serum levels of MMP-9.

To this end, in the current trial, effect of the prolongation of QRS duration over a certain period of time by short AVD permanent pacing on the circulating levels of a vascular extracellular matrix degradation marker, MMP-9, was examined.

ELIGIBILITY:
Inclusion Criteria:

* Normal LV systolic function (EF>50%),
* Healthy conduction systems
* Noncritical coronary stenoses or normal coronary arteries
* Ventricular pacing rate <10% in the last 6 months detected at the interrogation of the pacemakers

Exclusion Criteria:

* Intra-ventricular conduction abnormalities (baseline QRS >100 msec.),
* Mild to moderate aortic or mitral valve disease
* Presence of atrial fibrillation
* LV systolic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Change in MMP - 9 serum concentration from baseline to at the end of 3 weeks follow-up | 3 weeks
  MMP-9 serum concentration will be measured before and after short AV delay (wide QRS) pacing. Change in MMP-9 levels will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Department of Cardiology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided